CLINICAL TRIAL: NCT05470790
Title: Cross-Cultural Adaptation and Psychometric Properties Analysis of Arabic Version of Marx Activity Rating Scale and Knee Stability in Sports/Cutting-Pivoting Ability Scale for Saudi Athletes With Anterior Cruciate Ligament Injury
Brief Title: Arabic Version of Marx Activity Rating and Knee Stability in Sports/Cutting-Pivoting Ability Scales
Status: Recruiting | Type: Observational
Sponsor: Imam Abdulrahman Bin Faisal University (Other)
Collaborators: Qatif Central Hospital (Other)
Responsible Party: Principal Investigator, Majed Ali AlAbbad, Principal Investigator, Imam Abdulrahman Bin Faisal University
Other Study IDs: QCH-SREC0 4 /2022
Record Dates: First submitted 2022-07-20; First posted 2022-07-22 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Anterior Cruciate Ligament; Injuries
Keywords: Knee Injury; Sports Ability; Activity Level; Patient Report Outcome; Rating Scales
MeSH Terms: conditions — Wounds and Injuries; Knee Injuries | interventions — Patient Reported Outcome Measures

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- athletes with anterior cruciate ligament injuries
  Interventions: Other: patient reported outcome measures
- control
  Interventions: Other: patient reported outcome measures

INTERVENTIONS:
Other: patient reported outcome measures — Activity Rating Scale, Knee Stability in Sports/Cutting-Pivoting Ability scale, Knee Injury and Osteoarthritis Outcome Score, Lysholm Knee Score, and International Knee Documentation Committee Subjective Knee Form.

SUMMARY:
Anterior cruciate ligament (ACL) injuries are among the most common knee ligament injuries, causing joint instability and impairments. Besides being challenging, this type of injury greatly affects the athlete's passion and wellbeing, and it is associated with several risk factors. Injuries to the ACL are estimated to occur within 80,000 to 250,000 young, active and healthy athletes each year. This cross-sectional observational study aimed at translating, adapting cross-culturally, and investigating the psychometric properties of the Marx Activity Rating Scale (MARS) and the Knee Stability in Sports/Cutting-Pivoting Ability (KSS/CPA) scale in Saudi patients with anterior cruciate ligament injuries. For this study, a convenient sample size of 100 athletes with ACL injuries and healthy participants will be selected from different Saudi hospitals and clubs. Study participants will be informed about the study and a consent form will be obtained before they participate. A number of scales will be used as outcome measures, including the MARS, KSS/CPA scale, Knee Injury, and Osteoarthritis Outcome Score, Lysholm Knee Score, and International Knee Documentation Committee Subjective Knee Form. Internal consistency of both the MARS and KSS/CPA scales will be tested using Cronbach's alpha. A construct's validity will be measured by Spearman's correlation coefficient. Content validity can be determined by examining whether there are floor and ceiling effects. A significance level of 0.05 will be used to determine whether the data is significant. Ultimately, the study will help patients with ACL injuries to make informed decisions about their treatment, empower healthcare professionals to understand patients' concerns, and facilitate research.

ELIGIBILITY:
Inclusion Criteria:

1. An athlete with an orthopedic diagnosis of unilateral ACL injury
2. Age from 18 years to 45 years old
3. Participants who read and write in Arabic
4. Healthy participants that do not have lower limb injury limited participation in physical activity for at least six months.

Exclusion Criteria:

* 1 Patients with other lower limbs or different musculoskeletal injuries such as lower back pain may affect physical activity

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: sports population
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Arabic version of Marx activity rating scale | 1 minute
  The arabic version of Marx activity rating scale measures four activities: running, deceleration, cutting, and pivoting; higher scores indicate an increased frequency of knee-related activities. The frequency of performing these activities in the past 12 months is measured on a five-point scale. Based on the four items, the maximum score is 16 (if they answer "four or more times a week" for all four), and the minimum score is zero. For each item, one point will be awarded for each frequency category, beginning with "one time every month." and if participants answered "less than once a month" for one of the items, they will be awarded zero points; "once in a month," one point; "once a week," two points; etc.
Arabic version of knee stability in sports/cutting -pivoting ability scale | 1 minute
  The items in the Arabic version of knee stability in sports/cutting -pivoting ability scale are ranked on a Likert scale of 1 to 5, with response categories consisting of (A) normal, (B) near-normal, (C) abnormal, (D) severe abnormal, and (E) dysfunctional. knee stability in sports is a scale that emphasizes giving way to sensations and instability in the knees during linear activities (i.e., running in straight lines, accelerating, and decelerating), which involve lower-level motions. The cutting -pivoting ability scale section concerns the frequency, ability, and discomfort of performing pivotal activities. However, the ordinal knee stability in sports/cutting -pivoting ability scale will be converted into continuous variables (A = 100, B = 75, C = 50, D = 25, E = 0) and an overall self-assessment evaluation of knee function (0 = worst, 100 = best) will be recorded.

SECONDARY OUTCOMES:
Knee Injury and Osteoarthritis Outcome Score | 3 minutes
  There are five subscales with 42 items in the Knee Injury and Osteoarthritis Outcome Score questionnaire: Pain (9 items), Symptoms (7 items), Activities of Daily Living (17 items), Sport and Recreation (5 items), and Knee-related Quality of Life (QoL4). Each item wil be scored using a Likert scale ranging from 0 (no problem) to 4 (extreme problem). In addition, the subscale items will be rated on a scale of 0 to 100 using the following formula (100*average of subscale item scores/4*100), and higher scores indicate better health (100 = no knee problems) while low scores indicate poor health.
Lysholm Knee Score | 2 minutes
  Eight categories will be measured in the Lysholm Knee Score: instability (25 marks), pain (25 marks), catching (15 marks), stair climbing (10 marks), swelling (10 marks), need for support (5 marks), squatting (5 marks), and limping (5 marks). Each answer to the eight questions counts toward the total score, ranging from 0 to 100. High scores indicate better results and fewer symptoms. Lower scores indicate a problem with knee function.
International Knee Documentation Committee Subjective Knee Form | 2 minutes
  There are three main sections in the International Knee Documentation Committee Subjective Knee Form, overall consisting of 18 items: (1) symptoms (7 items), including swelling, pain, stiffness, giving way, and locking, (2) sports (1 item), (3) current knee function (9 items), and knee function after a knee injury (1 item) (not included in the overall score). The International Knee Documentation Committee Subjective Knee Form will be calculated by adding the scores of the individual items. The score will be then transformed into an overall score ranging from 0 to 100, with 100 indicating the absence of symptoms and higher levels of functioning. A total score of 100 will be calculated as (sum of items)/ (maximum possible score).

CONTACTS AND LOCATIONS:
Locations (1):
- Imam Abdulrahman Bin Faisal University, Dammam, Eastern Province, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared